CLINICAL TRIAL: NCT05805163
Title: A Culturally Relevant Communication and Support Plan to Ensure Access to and Use of Covid-19 Testing for Francophone African Born Immigrants
Brief Title: Tailored COVID-19 Testing Support Plan for Francophone African Born Immigrants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas Woman's University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: FY2023-241; R0704 (Other Grant/Funding Number: RADx-UP)
Record Dates: First submitted 2023-04-03; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: COVID19 Testing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants will be mailed a standard COVID-19 home-based test kit.
  Interventions: Behavioral: Standard COVID-19 home-based test kit
- Intervention (Experimental): Participants will be mailed a standard COVID-19 home-based test plus the FABI culturally sensitive COVID-19 educational pamphlet.
  Interventions: Behavioral: FABI tailored COVID-19 testing pamphlet; Behavioral: Standard COVID-19 home-based test kit

INTERVENTIONS:
Behavioral: FABI tailored COVID-19 testing pamphlet — FABI adapted COVID-19 educational pamphlet
  Arms: Intervention
Behavioral: Standard COVID-19 home-based test kit — Standard COVID-19 home-based test kit

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a culturally sensitive COVID-19 testing intervention designed for Francophone (French speaking) African Born Immigrants (FABI) . The main question this study aims to answer is whether or not a a culturally sensitive COVID-19 educational pamphlet added to the home-based test will improve testing rates compared to receiving a standard home-based test alone.

DETAILED DESCRIPTION:
Upon consenting, all participants will receive basic COVID-19 testing instructions from trained bilingual/bicultural Francophone African Born Immigrant (FABI) Community Health Workers (CHW's). Next, participants will be randomly assigned to either the control or intervention study arms. In the control condition (n=50) participants will receive a standard COVID-19 home-based test kit. In contrast, those assigned to the intervention condition (n=50) will receive the same COVID-19 home-based test kit plus a FABI culturally sensitive COVID-19 educational pamphlet. Lastly, (n=10) participants from each arm will be randomly selected to participate in qualitative interviews to assess their experiences with CHWs and their test kit.

ELIGIBILITY:
Inclusion Criteria: FABI living in Dallas Fort Worth (DFW) -

Exclusion Criteria: None

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Return rate | Tests returned within 3 months
  Ratio of returned tests over total tests provided

SECONDARY OUTCOMES:
Qualitative assessment | 2 months
  Qualitative assessment of experiences with CHWs, COVID-19 test kit, and FABI culturally sensitive COVID-19 educational pamphlet (if applicable)

IPD SHARING:
Plan to Share IPD: Undecided